CLINICAL TRIAL: NCT02291939
Title: Evaluation of Safety and Effectiveness of the FMwand Ferromagnetic Surgical System During Parotidectomy Surgery
Status: Completed | Type: Observational
Sponsor: Domain Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMT-IT-01
Record Dates: First submitted 2014-11-04; First posted 2014-11-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Parotid Diseases
MeSH Terms: conditions — Parotid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parotidectomy: Patients with an indication for surgical intervention for a parotidectomy.
  Interventions: Procedure: Parotidectomy

INTERVENTIONS:
Procedure: Parotidectomy — Surgical Intervention with the FMwand Surgical System

SUMMARY:
The objective of the clinical trial is to determine the suitability of the FMwand Ferromagnetic Surgical System for parotidectomy and Head & Neck surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for surgical intervention for a parotidectomy.
* ECOG status ≤ 2.
* Life expectancy > 3 months.
* Age ≥ 18 years old.
* Able to provide written informed consent and EU Data Protection Directive forms prior to admission to this study.
* Willingness to meet all of the expected requirements of this clinical protocol.

Exclusion Criteria:

* Age < 18 years old.
* Pregnant or breastfeeding.
* Vulnerable patient populations (homeless patients, patients with drug or alcohol dependence, etc.).
* Concomitant treatments that would affect clotting, post-operative healing, increased chances of infection.
* Previous radiation treatment
* Previous head or neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for surgical intervention for a parotidectomy.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative Serious Adverse Events as a Measure of Safety and Feasibility | 1 day after surgery
  Safety and feasibility will be assessed by evaluating intra-operative serious adverse events, if any, and their relationship with the FMwand Ferromagnetic Surgical System.

SECONDARY OUTCOMES:
Post-operative drainiage | Beginning day 2 after surgery and for the duration of hospital stay, an expected average of 6 days
  Evaluation of Post-operative Drainage
Swelling of surgical wound | Beginning day 2 after surgery and for the duration of hospital stay, an expected average of 6 days
  Evaluation of surgical wound appearance based on swelling
Necrosis of surgical margins | Beginning day 2 after surgery and for the duration of hospital stay, an expected average of 6 days
  Serosity and necrosis of margins
Length of hospital stay | Beginning day 2 after surgery and for the duration of hospital stay, an expected average of 6 days
  Number of days (post-operative) of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bellocchi, MD, Principal Investigator — San Camillo-Forlanini Hospital
Locations (1):
- San Camillo-Forlanini Hospital, Roma, Italy

REFERENCES:
- [Background] Bowers CA, Burns G, Salzman KL, McGill LD, Macdonald JD. Comparison of tissue effects in rabbit muscle of surgical dissection devices. Int J Surg. 2014;12(3):219-23. doi: 10.1016/j.ijsu.2013.12.014. Epub 2014 Jan 7. PMID 24406264
- [Background] Tok, S et al. Comparison of a Novel Thermal Surgical Technology with Monopolar and Carbon Dioxide Laser in a Rat Glioma Model. Poster presentation.
- [Background] MacDonald JD, Bowers CA, Chin SS, Burns G. Comparison of the effects of surgical dissection devices on the rabbit liver. Surg Today. 2014 Jun;44(6):1116-22. doi: 10.1007/s00595-013-0712-4. Epub 2013 Sep 5. PMID 24006128